CLINICAL TRIAL: NCT04700033
Title: Immersive Virtual Reality for Chronic Neuropathic Pain After Spinal Cord Injury: A Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, David Putrino, Director of Rehabilitation Innovation, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 18-0891
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Neuralgia; Spinal Cord Injuries; Chronic Pain
Keywords: Virtual Reality; Neuronal Plasticity; Neurological Rehabilitation; Immersive Virtual Reality
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries; Chronic Pain

STUDY DESIGN:
Intervention Model Description: The study is a single center, prospective randomized controlled clinical trial. The purpose of the study is to provide critical information about the efficacy of Immersive Virtual Reality (IVR) to decrease the experience of neuropathic pain in the upper and lower extremities of people with a spinal cord injury.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant, PI and Outcome Assessor remain blinded for the entirety of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Somatic IVR (Experimental): Participants with participate in Somatic IVR protocol three times per week for four weeks.
  Interventions: Device: Somatic IVR (sIVR)
- Distractive IVR (Active Comparator): Participants with participate in Distractive IVR protocol three times per week for four weeks.
  Interventions: Device: Distractive IVR (dIVR)
- Control IVR (Placebo Comparator): Participants with participate in Control IVR protocol three times per week for four weeks.
  Interventions: Device: Control IVR (cIVR)

INTERVENTIONS:
Device: Somatic IVR (sIVR) — This intervention will consist of an IVR protocol that is focused on somatic interaction that encourages disassociation between pain and visualization and movement of the affected limbs. Subjects in this group will be exposed to an IVR environment that cycles them through a series of stretching and mobility exercises for the affected limbs bilaterally.
  Arms: Somatic IVR
Device: Distractive IVR (dIVR) — This intervention will consist of an IVR that is focused on distracting the subject from the pain. Subjects in this group will be exposed to a variety of engaging landscape IVR environments, without the ability to visualize their own body.
  Arms: Distractive IVR
Device: Control IVR (cIVR) — This intervention will consist of an IVR exposure to a black screen for 20 minutes. No light, images or scenery will be present in the IVR and it will serve as a control condition for the trial.
  Arms: Control IVR

SUMMARY:
The aim of this study is to provide critical information about the efficacy of Immersive Virtual Reality (IVR) to decrease the experience of neuropathic pain in the upper and lower extremities of people with a spinal cord injury.

DETAILED DESCRIPTION:
When a spinal cord injury occurs, the spinal somatosensory circuit is thought to generate aberrant nociceptive impulses that the brain interprets as pain. Neuropathic pain (NP) affects 40 to 70% of people with SCI and is a very disabling clinical condition. Many treatment options have been offered, but provide limited effects, leaving people with SCI with a reduced quality of life. The study team believes that Immersive Virtual Reality (IVR) neurorehabilitation has the potential to be an effective treatment for chronic neuropathic pain. For this reason, the objective of this study is to evaluate the feasibility of using a virtual reality device to decrease chronic neuropathic pain in individuals with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury survivors (chronic only)
* Presence of neuropathic pain at or below SCI level for at least 6 months following trauma or disease of the spinal cord
* A pain intensity of at least 2 out of 10 in the numerical pain rating scale (NPRS) test at baseline
* Stable pharmacological treatment for at least 4 weeks prior to the study and throughout the trial

Exclusion Criteria:

* Psychiatric or other neurological disorders (Participants will not be excluded for having a SCI, if they score 0-30 points on the BDI, or if they report having anxiety)
* Head injuries causing cognitive or visual impairment
* Severe vertigo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Neuropathic Pain Symptom Inventory (NPSI) | Up to 10 Weeks
  Neuropathic Pain Symptom Inventory (NPSI): This scale was developed to assess both the quantitative and qualitative qualities of neuropathic pain (NP). It includes 12 items, assessing spontaneous pain, brief attacks of pain, provoked pain and abnormal sensations in the painful area. This is a sensitive tool for measuring changes in neuropathic pain after a therapeutic intervention. Total score range for NPSI is 0-100, higher scores indicate more severity.

SECONDARY OUTCOMES:
User Experience Score (UES) | 14 Days
  Participants rate their experience using the technology on a scale with a total score range of 0 to 10, where 0 means no enjoyment and 10 means very high levels of enjoyment.
Spinal Cord Independence Measure (SCIM III) | Up to 10 Weeks
  Spinal cord independence measure (SCIM III) measures the ability of patients with SCI to perform everyday tasks. SCIM is used for quantitative functional outcome assessment following interventions designed to promote recovery from spinal cord injury and to increase functional achievement; it covers 19 tasks in 16 categories, with a score range 0-100; all activities of daily living, grouped into four areas of function (subscales): Self-Care (scored 0-20), Respiration and Sphincter Management (0-40), Mobility in Room and Toilet (0-10), and Mobility Indoors and Outdoors (0-30). VR neurorehabilitation has shown to improve motor function as well as to reduce neuropathic pain in incomplete SCI patients. The study team is planning to monitor the effects that this IVR protocol has in motor recovery. Total score range for SCIM II is 0 - 100, where a score of 0 defines total dependence and a score of 100 is indicative of complete independence.
Numerical Pain Rating Scale (NPRS) | 16 Days
  Users report the score of both neuropathic and other pain. The total score range is from 0 to 10, lowest score indicating 0, "No pain" and highest score indicating 10, "Pain as bad as it could be". The type of "other" pain will also be recorded (musculoskeletal, etc).
Beck Depression Inventory (BDI) | Up to 10 Weeks
  Beck Depression Inventory (BDI): Depression symptoms are estimated to be highly prevalent in SCI population and are associated with a myriad of negative outcomes including lower functional independence, and greater incidence of pain. This questionnaire is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. Depression may be a major contributor to a lack of reduction of pain, the study team expects subjects with high BDI score may have worse results after the IVR. Total score range for BDI is 0 - 63; scores from 0 through 9 indicate no or minimal depression; from 10 through 18 indicate mild to moderate depression; from 19 through 29 indicate moderate to severe depression; and from 30 through 63 indicate severe depression.
Patient's Global Impression of Change (PGIC) | Up to 10 Weeks
  Self-reported relieving effect: At the end of the treatment (post-intervention), the Patient's Global Impression of Change (PGIC) will evaluate both motor function and pain. The total score range includes no change (score 0-1), minimally improved (score 2-3), much improved (score 4-5), and very much improved (score 6-7) as the highest score. The patients will answer the following question: "Since beginning treatment at this program, how would you describe the change (if any) in activity limitations, symptoms, emotions, and overall quality of life related to your condition?".
Immersive Tendencies Questionnaire (ITQ) | Up to 10 Weeks
  Immersive tendencies questionnaire (ITQ): In the field of virtual reality, presence and immersion are standard measures of an individual's sense of engagement and involvement in an activity. The study team expects that high levels of immersion might indicate greater engagement and therefore reduction of the pain. Total score range for ITQ: 18 - 126.
UQO- Presence Questionnaire (UPO-PQ) | 16 Days
  The UQO Presence questionnaire (UQO-PQ): Presence can be a major factor that determines the quality and success of a virtual environment implementation. Several factors such as impression of being present, realness, and discomfort are measured in this questionnaire. The questionnaire has users rank the extent the agree with each question with the total score range of 0 - 100; the lowest score indicating 0 - "Not at all" and the highest score indicating 100- "Totally".
Neuropathic Pain Scale (NPS) | Up to 10 Weeks
  Neuropathic Pain Scale (NPS): This scale was developed to assess both the quantitative and qualitative qualities of neuropathic pain (NP). It includes 11 items, assessing global pain intensity, unpleasantness, and one item which allows the patient to describe the temporal aspects of their pain and its qualities in their own words.The remaining 8 items assess specific NP qualities: "Sharp," "Hot," "Dull," "Cold," "Sensitive," "Itchy," "Deep," and "Surface." This is a sensitive tool for measuring changes in neuropathic pain after a therapeutic intervention. Total score range for NPS is 0 - 100, higher scores indicate more severity.

CONTACTS AND LOCATIONS:
Overall Officials: David Putrino, PT, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No